CLINICAL TRIAL: NCT01058655
Title: A Phase I/II Study of RAD001 and AV-951 in Patients With Refractory, Metastatic Colorectal Cancer
Brief Title: RAD001 and AV-951 in Patients With Refractory, Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Novartis (Industry); AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Brian Wolpin, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-276
Record Dates: First submitted 2009-10-29; First posted 2010-01-29 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-02

CONDITIONS: Gastrointestinal Cancer
Keywords: Colorectal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms | interventions — Everolimus; tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase I Cohort 1: Everolimus 5 mg + Tivozanib 1 mg (Experimental): Patients received oral everolimus daily continuously and oral tivozanib daily for 3 of a 4 weeks cycle. Patients are treated until disease progression, unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Everolimus; Drug: Tivozanib
- Phase I Cohort 2: Everolimus 10 mg + Tivozanib 1 mg (Experimental): Patients received oral everolimus daily continuously and oral tivozanib daily for 3 of a 4 weeks cycle. Patients are treated until disease progression, unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Everolimus; Drug: Tivozanib
- Phase I Cohort 3: Everolimus 10 mg + Tivozanib 1.5 mg (Experimental): Patients received oral everolimus daily continuously and oral tivozanib daily for 3 of a 4 weeks cycle. Patients are treated until disease progression, unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Everolimus; Drug: Tivozanib
- Phase II: Everolimus 10 mg + Tivozanib 1 mg (Experimental): Patients received oral everolimus daily continuously and oral tivozanib daily for 3 of a 4 weeks cycle. Patients are treated until disease progression, unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Everolimus; Drug: Tivozanib

INTERVENTIONS:
Drug: Everolimus
  Other Names: RAD001; Afinitor
Drug: Tivozanib
  Other Names: AV-951

SUMMARY:
Research has shown that anti-angiogenic agents can be effective therapies to treat cancer. Anti-angiogenic agents target the blood vessels required for tumors to grow. Vascular endothelial growth factor (VEGF) is one of the cell pathways used for this blood vessel growth. When the investigators interfere with the VEGF pathway, the investigators inhibit this blood vessel growth which is required by tumors. One of the study drugs being used, tivozanib (AV-951), selectively interferes with the VEGF pathway. The second study drug being used, everolimus (RAD001) interferes with the mTOR pathway. The mTOR pathway is another pathway involved in blood vessel and tumor cell growth. By combining these two drugs the investigators hope to slow or reverse tumor cell growth in patients whose tumors have become resistant to other therapies for their disease.

DETAILED DESCRIPTION:
Primary Objective

Phase I

* To determine the safety, tolerability, and maximally tolerated dose (MTD) of everolimus and tivozanib administered in combination to patients with advanced gastrointestinal tumors.

Phase II

* At the MTD, to assess progression-free survival associated with everolimus and tivozanib in patients with refractory, metastatic colorectal cancer.

Secondary Objectives

Phase II

* To assess tumor response rate.
* To assess overall survival.

ELIGIBILITY:
For the Phase I component:

Inclusion Criteria:

* 18 years of age or older
* Histologic confirmation of a gastrointestinal malignancy, limited to cancer of the esophagus, stomach, small bowel, liver, biliary tract, gallbladder, pancreas, large bowel, appendix, rectum and anus.
* Locally advanced or metastatic disease
* Disease that: a) has recurred or progressed following standard therapy, b) for which no standard therapy currently exists, or c) for which the subject is not a candidate for or unwilling to undergo standard therapy. There is no limit to the number of prior regimens received by the patient.
* ECOG Performance Status of 0, 1 or 2
* Life expectancy of at least 12 weeks
* Adequate organ function as outlined in the protocol
* At least 4 weeks is required from : a) previous regimen of chemotherapy, b) immunotherapy or biological therapy, c) other investigational agents, and d) radiotherapy.
* At least 4 weeks is required from treatment of bevacizumab
* At least 4 weeks is required from prior systemic hormonal therapy or treatment with strong CYP3A4 inducers or inhibitors
* If female and of child bearing potential, documentation of negative pregnancy test prior to enrollment.

Exclusion Criteria:

* Prior therapy with inhibitors of mTOR or VEGFR (prior treatment with bevacizumab is allowed).
* Clinically apparent CNS metastases or carcinomatous meningitis
* Clinically significant cardiovascular disease
* Major surgery within 4 weeks of the start of study treatment or patients who have not recovered from the side effects of any major surgery.
* Active bleeding diathesis or history of Grade 2 or greater clinically significant bleeding within 3 months of enrollment
* Active infection requiring antibiotics
* Participants with a known positive history of chronic Hepatitis B viral infection or known positive HBV-DNA test are excluded.
* History of interstitial pneumonitis or severely impaired lung function defined as 88% or less O2 saturation at rest in room air
* Immunocompromise or chronic use of immunosuppressant medications
* Uncontrolled serious medical or psychiatric illness
* Subjects with non-healing wounds, active peptic ulcers, or unhealed bone fractures
* Significant proteinuria, defined as urine dipstick protein of 3+ or greater
* Concurrent malignancy (other than non-melanoma skin cancer) diagnosed within the past 3 years or any currently active malignancy
* Elevated fasting levels of the following: serum cholesterol, serum triglycerides, and serum glucose
* Patients who are pregnant or lactating
* Malabsorption, uncontrolled vomiting or diarrhea, or any disease significantly affecting gastrointestinal function that could interfere with absorption of study drugs
* Inability to swallow pills

For the phase II component, only patients with metastatic colorectal cancer will be enrolled.

For the Phase II component:

Inclusion Criteria (Phase II):

* 18 years of age or older
* Histologic confirmation of colorectal cancer
* Stage IV disease
* At least one site of disease measurable by RECIST criteria
* Receipt of or intolerance to a fluoropyrimidine (fluorouracil or capecitabine), irinotecan, oxaliplatin, bevacizumab, and a monoclonal antibody to epidermal growth factor receptor (cetuximab or panitumumab). If a patient's tumor was K-RAS mutation positive, then previous treatment with cetuximab or panitumumab is not required.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Life expectancy of at least 12 weeks
* Adequate organ function as outlined in the protocol
* At least 3 weeks is required from: (a) previous regimen of chemotherapy, (b)immunotherapy or biological therapy, (c) other investigational agents, and (d) radiotherapy. Of note, concomitant radiotherapy is NOT allowed, while a patient is on protocol.
* At least 3 weeks is required from prior treatment with bevacizumab
* At least 3 weeks is required since prior systemic hormonal therapy or treatment with strong CYP3A4 inducers or inhibitors.
* Negative pregnancy test for women of child bearing potential

Exclusion Criteria (Phase II):

* Prior therapy with inhibitors of mTOR or VEGFR (prior treatment with bevacizumab is allowed)
* Clinically apparent CNS metastases or carcinomatous meningitis, as determined by physical examination and imaging studies
* Clinically significant cardiovascular disease, defined as follows:

(A)Symptomatic congestive heart failure, (B)Symptomatic coronary artery disease or myocardial infarction within 3 months of enrollment, (C)Cardiac arrhythmias not controlled with medication, (D)Deep venous thrombosis or pulmonary embolus within the last 6 months, (E) Cerebrovascular accident within the last 12 months, (F)Poorly controlled hypertension, defined as systolic pressure > 150 mmHg or diastolic pressure > 100 mmHg documented on 2 consecutive measurements taken at least 24 hours apart, (G)Symptomatic peripheral vascular disease, defined as claudication on walking ≤

1 block

* Major surgery within 4 weeks of the start of study treatment or patients who have not recovered from the side effects of any major surgery. Major surgery defined as those surgeries that require general anesthesia
* Active bleeding diathesis or history of grade 2 or higher clinically significant bleeding (hemoptysis, hematemesis, hematochezia, or melena) within 3 months of enrollment
* Active infection requiring antibiotics
* Participants with a known positive history of chronic Hepatitis B viral infection or known positive HBV-DNA test are excluded.
* History of interstitial pneumonitis or severely impaired lung function defined as less than or equal to 88% O2 saturation at rest in room air.
* Immunocompromise or chronic use of immunosuppressant medications (prednisone ≤ 10 mg daily or the equivalent of a comparable steroid is allowed, if deemed necessary by a study investigator)
* Uncontrolled serious medical or psychiatric illness
* Subjects with non-healing wounds, active peptic ulcers, or unhealed bone fractures
* Significant proteinuria, defined as urine dipstick protein 3+ or greater
* Concurrent malignancy (other than non-melanoma skin cancer) diagnosed within the past 3 years or any currently active malignancy.
* Elevated fasting levels of the following: serum cholesterol, serum triglycerides, and serum glucose.
* Patients who are pregnant or lactating
* Malabsorption, uncontrolled vomiting or diarrhea, or any disease significantly affecting gastrointestinal function that could interfere with absorption of study drugs
* Inability to swallow pills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-02; Primary Completion 2013-09 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Wolpin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wolpin BM, Ng K, Zhu AX, Abrams T, Enzinger PC, McCleary NJ, Schrag D, Kwak EL, Allen JN, Bhargava P, Chan JA, Goessling W, Blaszkowsky LS, Supko JG, Elliot M, Sato K, Regan E, Meyerhardt JA, Fuchs CS. Multicenter phase II study of tivozanib (AV-951) and everolimus (RAD001) for patients with refractory, metastatic colorectal cancer. Oncologist. 2013;18(4):377-8. doi: 10.1634/theoncologist.2012-0378. Epub 2013 Apr 11. PMID 23580238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from February 2010 through June 2011.
Period: Overall Study
Arm/Group | Phase I Cohort 1: Everolimus 5 mg + Tivozanib 1 mg | Phase I Cohort 2: Everolimus 10 mg + Tivozanib 1 mg | Phase I Cohort 3: Everolimus 10 mg + Tivozanib 1.5 mg | Phase II: Everolimus 10 mg + Tivozanib 1 mg
Started | 3 | 3 | 8 | 42
Evaluable | 3 | 3 | 6 | 40
Completed (Since treatment was not of fixed duration, all participants were considered as 'Not Completed'.) | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 8 | 42
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 4
Not completed — Prolonged Treatment Delay | 0 | 0 | 0 | 2
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 1
Not completed — Clinical Progression (non-RECIST) | 1 | 0 | 0 | 7
Not completed — Death | 0 | 1 | 1 | 0
Not completed — Disease Progression | 1 | 2 | 4 | 24
Not completed — Other | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled patients.
Groups:
- Phase I Cohort 1: Everolimus 5 mg + Tivozanib 1 mg; Phase I Cohort 2: Everolimus 10 mg + Tivozanib 1 mg; Phase I Cohort 3: Everolimus 10 mg + Tivozanib 1.5 mg; Phase II: Everolimus 10 mg + Tivozanib 1 mg: Patients received oral everolimus daily continuously and oral tivozanib daily for 3 of the 4 week cycle. Patients are treated until disease progression, unacceptable toxicity or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Phase I Cohort 1: Everolimus 5 mg + Tivozanib 1 mg | Phase I Cohort 2: Everolimus 10 mg + Tivozanib 1 mg | Phase I Cohort 3: Everolimus 10 mg + Tivozanib 1.5 mg | Phase II: Everolimus 10 mg + Tivozanib 1 mg | Total
Number analyzed (Participants) | 3 | 3 | 8 | 42 | 56
Age, Continuous [Median (Full Range); unit: years] | 58 [50 to 70] | 47 [40 to 68] | 63 [48 to 82] | 56 [36 to 82] | 59 [36 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 3 | 23 | 28
  Male | 3 | 1 | 5 | 19 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2 | 4
  White | 2 | 3 | 7 | 38 | 50
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 8 | 42 | 56

OUTCOME MEASURES:

1. Primary Outcome: Everolimus Maximum Tolerated Dose (MTD) [Phase I]
Description: The everolimus MTD in combination with tivozanib is determined by the number of patients who experience a dose limiting toxicity (DLT). See subsequent primary outcome measure for the DLT definition. The MTD is defined as the highest dose at which fewer than one-third of patients experience a DLT. If no DLTs are observed, the MTD is not reached.
Time Frame: Patients were assessed continuously for toxicity while on study. The observation period for MTD evaluation was the first 28 days (cycle 1) of treatment.
Population: All PI patients who received at least one dose of the study drug were evaluable for MTD unless patient withdrew before completing 1 cycle of therapy for reason other than dose-limiting toxicity.
Measure: Number; unit: mg daily for 4 weeks of a 4 week cycle
Groups:
- Phase I: Evaluable: All phase I patients received oral everolimus daily continuously and oral tivozanib daily for 3 of a 4 weeks cycle according to the established dose escalation schedule. Patients who withdrew before completing 1 cycle of therapy for reason other than dose-limiting toxicity were not evaluable and replaced.
Arm/Group | Phase I: Evaluable
Number analyzed (Participants) | 12
mg daily for 4 weeks of a 4 week cycle | 10

2. Primary Outcome: Tivozanib Maximum Tolerated Dose (MTD) [Phase I]
Description: The tivozanib MTD in combination with everolimus is determined by the number of patients who experience a dose limiting toxicity (DLT). See subsequent primary outcome measure for the DLT definition. The MTD is defined as the highest dose at which fewer than one-third of patients experience a DLT. If no DLTs are observed, the MTD is not reached.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: mg daily for 3 weeks of a 4 week cycle
Arm/Group | Phase I: Evaluable
Number analyzed (Participants) | 12
mg daily for 3 weeks of a 4 week cycle | 1.0

3. Primary Outcome: Dose Limiting Toxicity (DLT) [Phase I]
Description: A DLT was defined as a treatment-related (attribution possible, probable, definite) adverse event that meets any of the following criteria: Grade 3 (G3) or higher non-hematologic toxicity (excluding, nausea, vomiting, diarrhea, alopecia, hypertension, hypercholesterolemia, or hypertriglyceridemia); G3 diarrhea, nausea or vomiting lasting > 48 hours or leading to hospitalization, despite aggressive anti-diarrheal or anti-emetic medications; G4 diarrhea, despite aggressive anti-diarrheal medications; G4 vomiting, despite aggressive anti-emetic medications; G3 hypertension, for which blood pressure cannot be reduced to <150/100 with anti-hypertensive therapies; G4 hypertension or severe hypertension, as defined by systolic blood pressure >180 mmHg or diastolic blood pressure > 110 mmHg; G4 hypercholesterolemia or hypertriglyceridemia lasting > 7 days, despite appropriate use of anti-hyperlipidemic medications; G4 hematologic toxicity lasting for >5 days, including leukopenia, neutropen
Time Frame: Patients were assessed continuously for toxicity while on study. The observation period for DLT evaluation was the first 28 days (cycle 1) of treatment.
Population: All PI patients who received at least one dose of the study drug were evaluable for DLT. The 2 DLTs experienced by participants in dose level cohort 3 were grade 3 fatigue and dehydration.
Measure: Number; unit: Participants with DLT
Arm/Group | Phase I Cohort 1: Everolimus 5 mg + Tivozanib 1 mg | Phase I Cohort 2: Everolimus 10 mg + Tivozanib 1 mg | Phase I Cohort 3: Everolimus 10 mg + Tivozanib 1.5 mg
Number analyzed (Participants) | 3 | 3 | 6
Participants with DLT | 0 | 0 | 2

4. Primary Outcome: Progression-Free Survival (PFS) [Phase II]
Description: PFS based on the Kaplan-Meier method is defined as the time from study entry to the earliest documentation of disease progression (PD) or death. Participants alive without evidence of PD were censored at the earliest date of last disease assessment. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was assessed radiographically to document clinical progression every 2 cycles on treatment. Participants were followed for up to 16 months since study entry.
Population: The analysis dataset is comprised of all evaluable phase II patients.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase II: Everolimus 10 mg + Tivozanib 1 mg [Evaluable]: Patients received oral everolimus daily continuously and oral tivozanib daily for 3 of the 4 week cycle. Patients are treated until disease progression, unacceptable toxicity or withdrawal of consent.
Arm/Group | Phase II: Everolimus 10 mg + Tivozanib 1 mg [Evaluable]
Number analyzed (Participants) | 40
months | 3.0 [1.9 to 3.6]

5. Secondary Outcome: Disease Control Rate (DCR) [Phase II]
Description: Disease Control Rate is defined as the percentage of patients who achieve confirmed stable disease (SD) or better on treatment based on RECIST 1.0 criteria. Per RECIST 1.0 for target lesions, complete response (CR) is disappearance of all target lesions and partial response (PR) is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. Progressive disease (PD) is at least a 20% increase in sum LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started. SD is neither PR nor PD. For non-target lesions, PD is the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Disease was assessed every 2 cycles on treatment. Median treatment duration on this study cohort was 2 months (range 1-16).
Population: The analysis dataset is comprised of all evaluable phase II patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: Everolimus 10 mg + Tivozanib 1 mg [Evaluable]
Number analyzed (Participants) | 40
percentage of participants | 50 [34 to 66]

6. Secondary Outcome: Overall Survival (OS) [Phase II]
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or date last known alive.
Time Frame: Long-term follow-up for survival was not specified per protocol. Participants were followed for up to 20 months on this study.
Population: The analysis dataset is comprised of all evaluable phase II patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Everolimus 10 mg + Tivozanib 1 mg [Evaluable]
Number analyzed (Participants) | 40
months | 5.6 [4.4 to 10.6]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed continuously throughout treatment. Treatment duration was a median of 2 months (range 1-16 months) in this study cohort.
Description: AEs with treatment-attribution of possibly, probably or definitely were classified as serious if maximum grade 3-5 or other if grade 1-2 per CTCAEv3.
Arm/Group | Phase I Cohort 1: Everolimus 5 mg + Tivozanib 1 mg | Phase I Cohort 2: Everolimus 10 mg + Tivozanib 1 mg | Phase I Cohort 3: Everolimus 10 mg + Tivozanib 1.5 mg | Phase II: Everolimus 10 mg + Tivozanib 1 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/8 | 5/42
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 3/8 | 30/42
Other Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 6/8 | 32/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Cohort 1: Everolimus 5 mg + Tivozanib 1 mg (N=3) | Phase I Cohort 2: Everolimus 10 mg + Tivozanib 1 mg (N=3) | Phase I Cohort 3: Everolimus 10 mg + Tivozanib 1.5 mg (N=8) | Phase II: Everolimus 10 mg + Tivozanib 1 mg (N=42)
ALT- SGPT (Investigations) | 0 | 0 | 0 | 1
AST- SGOT (Investigations) | 0 | 0 | 0 | 5
Abdomen- pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Alkaline phosphatase (Investigations) | 0 | 0 | 2 | 2
Back- pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bilirubin (Investigations) | 0 | 0 | 0 | 2
Breast- pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Chest wall- pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Chest/thoracic pain NOS (General disorders) | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Creatinine (Investigations) | 0 | 0 | 0 | 1
Death - disease progression NOS (General disorders) | 0 | 0 | 0 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 0 | 0 | 0 | 6
Fatigue (General disorders) | 0 | 0 | 1 | 5
Head/headache (Nervous system disorders) | 0 | 0 | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 3
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 11
Infection w/ unk ANC kidney (Infections and infestations) | 0 | 0 | 0 | 1
Intra-op injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Intra-op injury Colon (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Intra-op injury Spinal cord (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lymphopenia (Investigations) | 0 | 0 | 0 | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Muco/stomatitis by exam- oral cavity (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Neutrophils (Investigations) | 0 | 0 | 0 | 2
Obstruction- small bowel NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Platelets (Investigations) | 0 | 0 | 0 | 10
Rectum- pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0
Stenosis (incl anastomotic) biliary tree (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Varices (esophageal)- hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Cohort 1: Everolimus 5 mg + Tivozanib 1 mg (N=3) | Phase I Cohort 2: Everolimus 10 mg + Tivozanib 1 mg (N=3) | Phase I Cohort 3: Everolimus 10 mg + Tivozanib 1.5 mg (N=8) | Phase II: Everolimus 10 mg + Tivozanib 1 mg (N=42)
ALT- SGPT (Investigations) | 1 | 0 | 2 | 7
AST- SGOT (Investigations) | 3 | 0 | 1 | 17
Abdomen- pain (Gastrointestinal disorders) | 1 | 1 | 0 | 15
Alkaline phosphatase (Investigations) | 0 | 0 | 0 | 16
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 11
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Ascites (non-malignant) (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Atrial tachycardia/PAT (Cardiac disorders) | 0 | 0 | 0 | 1
Back- pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 6
Bilirubin (Investigations) | 0 | 1 | 0 | 4
Bone- pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Bronchospasm- wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Chest wall- pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
CNS- hemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 6
Creatinine (Investigations) | 0 | 0 | 0 | 5
Cystitis (Renal and urinary disorders) | 0 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dental/teeth/peridontal- pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 2 | 1 | 4 | 13
Distention/bloating- abdominal (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 6
Edema head and neck (General disorders) | 0 | 0 | 0 | 1
Edema limb (General disorders) | 1 | 1 | 1 | 4
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
External ear- pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Extremity-lower (gait/walking) (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 3 | 17
Fever w/o neutropenia (General disorders) | 0 | 0 | 0 | 3
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Head/headache (Nervous system disorders) | 1 | 0 | 0 | 6
Hematoma (Vascular disorders) | 0 | 0 | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 1 | 1 | 1 | 20
Hemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 13
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 18
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 3 | 0 | 3 | 17
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 15
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 19
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 16
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 14
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0 | 3 | 7
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2
Infection Gr0-2 neut- bronchus (Infections and infestations) | 0 | 0 | 0 | 1
Infection Gr0-2 neut- dental-tooth (Infections and infestations) | 0 | 0 | 0 | 1
Infection Gr0-2 neut- oral cavity (Infections and infestations) | 0 | 0 | 0 | 1
Infection Gr0-2 neut- sinus (Infections and infestations) | 0 | 0 | 0 | 1
Infection Gr0-2 neut- urinary tract (Infections and infestations) | 0 | 0 | 0 | 3
Infection w/ unk ANC bronchus (Infections and infestations) | 0 | 0 | 0 | 1
Infection w/ unk ANC vagina (Infections and infestations) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1
Joint- pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Leukocytes (Investigations) | 0 | 0 | 0 | 4
Lip- pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lymph node- pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphopenia (Investigations) | 0 | 0 | 0 | 1
Mental status (Nervous system disorders) | 0 | 0 | 0 | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 2 | 1 | 2 | 7
Muco/stomatitis by exam- oral cavity (Gastrointestinal disorders) | 0 | 0 | 0 | 9
Muscle- pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 14
Neck- pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neutrophils (Investigations) | 1 | 0 | 0 | 9
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Nose- hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Pelvic- pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Platelets (Investigations) | 1 | 0 | 4 | 16
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 7
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 7
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 5
Rectum- pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0
Rigors/chills (General disorders) | 0 | 0 | 0 | 2
Stenosis (incl anastomotic) duodenum (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomach- pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Throat/pharynx/larynx- pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 0 | 0 | 2
Urethra- pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 0 | 0 | 3
Urinary hemorrhage NOS (Renal and urinary disorders) | 0 | 0 | 0 | 1
Vaginal discharge (non-infectious (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 5
Weight loss (Investigations) | 1 | 1 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No